CLINICAL TRIAL: NCT00869375
Title: Use of Clearway™ Balloon vs. Mechanical Thrombectomy as Initial Treatment for Acute Limb Ischemia: A Randomized Controlled Trial
Brief Title: Use of Clearway™ Balloon vs. Mechanical Thrombectomy as Initial Treatment for Acute Limb Ischemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: very low enrollment due to low access to study population
Sponsor: University of Oklahoma (Other)
Collaborators: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEARWAY-CLI
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Critical Limb Ischemia
Keywords: acute or critical limb ischemia with angiographic thrombus
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLEARWAY GROUP (Active Comparator): Endovascular peripheral intervention - Percutaneous transluminal angioplasty with simultaneous in situ thrombolysis (local thrombolytic plus low pressure balloon angioplasty) with Clearway balloon
  Interventions: Device: Endovascular peripheral intervention
- ANGIOJET GROUP (Active Comparator): Endovascular peripheral intervention - Percutaneous transluminal angioplasty with simultaneous mechanical thrombectomy with AngioJet Rheolytic Thrombectomy System
  Interventions: Device: Endovascular peripheral intervention

INTERVENTIONS:
Device: Endovascular peripheral intervention — Clearway Balloon: percutaneous transluminal angioplasty with simultaneous in situ thrombolysis using the Clearway balloon AngioJet Rheolytic Thrombectomy System: percutaneous transluminal angioplasty with simultaneous mechanical thrombectomy using the Angiojet
  Other Names: Clearway Balloon; AngioJet Rheolytic Thrombectomy System

SUMMARY:
The purpose of this study is to compare the effects (positive and negative) of two different devices available to treat people with critical limb ischemia, which involves a sudden decrease in blood flow to the leg that causes a potential threat to the limb and causes pain at rest, ulcers or gangrene.

One device is the Clearway balloon, which delivers a drug to dissolve the clot where the blockage is. The other device is the Angiojet, which removes the clot in a mechanical way ("vacuum" effect). This research is being done because currently there is no single proven effective treatment for this condition. Even though, both these devices are commonly used in the clinical practice to treat critical limb ischemia, there are no studies that compare these devices and help us see which one may be better for these patients.

DETAILED DESCRIPTION:
This prospective randomized clinical trial in patients with peripheral vascular disease and acute or subacute arterial thrombosis will compare percutaneous transluminal angioplasty and simultaneous in situ thrombolysis using the Clearway balloon system with mechanical thrombectomy with the Angiojet system. Main endpoints are the time to successful revascularization, the frequency of distal embolization and the incidence of bleeding complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 85 years of age
* Diagnosis of acute limb ischemia (defined as an abrupt onset of lower extremity pain with loss of peripheral pulses and absent Doppler pulses in at least one artery and/or ultrasonographic evidence of decreased or absent blood flow to the affected limb) or Diagnosis of critical limb ischemia (defined as resting lower extremity pain with an ABI of <0.4 and/or ultrasonographic evidence of decreased or absent blood flow to the affected limb).
* Angiographic confirmation of thrombus.
* Need of an intervention within 21 days of the onset of symptoms

Exclusion Criteria:

* Any contraindication for thrombolytic therapy

ABSOLUTE CONTRAINDICATIONS:

A. Any history of intracranial hemorrhage; recent (within three months) hemorrhagic cerebrovascular accident (CVA) / transient ischemic attack (TIA) or significant closed head or facial injury.

B. Known intracranial neoplasm or arteriovenous malformation. C. Suspected aortic dissection. D. Active bleeding diathesis or hemostatic defects: (Excluding menses); active internal

RELATIVE CONTRAINDICATIONS:

Fibrinolytic therapy may be used with the presence of these conditions upon clinical assessment or treatment dependent upon bleeding risks:

A. History of chronic, severe, and poorly controlled blood pressure or Severe uncontrolled hypertension on presentation (SBP >180, DBP >110).

B. History of prior ischemic stroke (greater than 3 months) dementia, or known intracranial pathology not covered in absolute contraindications.

C. Traumatic or prolonged CPR (> 10 minutes), major surgery (< 3 weeks), or recent trauma, including head trauma (2-4 weeks).

D. Recent (within 2 to 4 weeks) internal bleeding. E. Noncompressible vascular punctures. F. Pregnancy or recent obstetrical delivery. G. Active peptic ulcer disease. H. Anticoagulant use (INR > 2-3)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Emilio Exaire, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CLEARWAY GROUP; ANGIOJET GROUP: 3 patients were randomized in this group.
Period: Overall Study
Arm/Group | CLEARWAY GROUP | ANGIOJET GROUP
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLEARWAY GROUP | ANGIOJET GROUP | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 45 [42 to 49] | 63 [57 to 74] | 54 [42 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Diabetes [Number; unit: participants] | 2 | 1 | 3
Hypertension [Number; unit: participants] | 2 | 2 | 4
Dyslipidemia [Number; unit: participants] | 2 | 1 | 3
Current smokers [Number; unit: participants] | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Immediate Distal Embolization Detected by Angiographic and/or Clinical Evidence
Time Frame: 24 hours after the procedure
Measure: Number; unit: participants
Groups:
- CLEARWAY GROUP; ANGIOJET GROUP: No patients had distal embolization
Arm/Group | CLEARWAY GROUP | ANGIOJET GROUP
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

2. Primary Outcome: Incidence of Bleeding Complications
Time Frame: 24 hours after the procedure
Measure: Number; unit: participants
Groups:
- CLEARWAY GROUP: 4 patients were randomized in this group. One patient was excluded since intervention was not required.
Arm/Group | CLEARWAY GROUP | ANGIOJET GROUP
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | CLEARWAY GROUP | ANGIOJET GROUP
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLEARWAY GROUP (N=3) | ANGIOJET GROUP (N=3)
Emergency surgery (Vascular disorders) | 1 (1) | 0 (0) — One patient in the clearway group required emergency embolectomy due to failure to revascularize. This was not deemed to be secondary to a failure of strategy or failure of device but rather to the severity and extension of the thrombbus.

LIMITATIONS AND CAVEATS:
The main limitation of this trial was slow enrollment. This led to early termination leading to small numbers of subjects analyzed. This makes the results uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No